CLINICAL TRIAL: NCT00188305
Title: A Randomized Trial of Cancer Risk and Health Education in Relatives of Colorectal Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: UHN04-0729-CE
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Colon Cancer; Colonic Neoplasms
Keywords: Risk counselling; Health education; Prevention; Behavioral; Screening; Intervention; Telephone vs in person
MeSH Terms: conditions — Colonic Neoplasms; Health Education; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 In person (Experimental): In person general health, colorectal cancer risk information and screening recommendations.
  Interventions: Behavioral: General health counselling and risk information
- 2 Telephone (Active Comparator): Telephone general health counselling, colorectal cancer risk information and screening recommendations.
  Interventions: Behavioral: General health counselling and risk information
- 3 Control (Placebo Comparator): Standard care for 2 months followed by summary letter with general health information, colorectal cancer risk information and screening recommendations.
  Interventions: Behavioral: General health counselling and risk information

INTERVENTIONS:
Behavioral: General health counselling and risk information — General health counselling and risk information

SUMMARY:
Having at least one first-degree relative (FDR) with colon cancer increases an individual's risk of developing the disease. Many relatives of cancer patients are ineligible for genetic testing and, therefore, do not receive information from a healthcare provider about the disease. Providing relatives of cancer patients with information about their risk of developing colon cancer, screening information, and other colon-related health information, may increase knowledge and screening compliance as has been shown in relatives of breast cancer patients. The primary aim of this study is to test the efficacy of two modes (in-person vs. telephone) of providing a risk counseling and health promotion intervention for relatives of cancer patients on measures of knowledge of colon cancer risk and health-related factors, comprehension of risk, understanding of screening recommendations and intent to adopt an appropriate screening regimen. Participants will be randomized into one of three study arms (in-person, telephone, control). An assessment pre- and post- intervention will be conducted. In addition, longer-term follow-ups will be carried out two months and one year following the intervention to examine the sustainability of the intervention effect.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer death in North America, despite being referred to as preventable and curable if detected early. Early detection through preventive screening has been found to decrease CRC death. However, adherence to CRC screening is poor, both in average risk and higher risk individuals. Lack of knowledge of CRC risk and screening recommendations, and psychological factors, such as perceived risk of CRC have been cited as important factors associated with screening compliance. By increasing knowledge and appropriate risk comprehension, it is possible to increase lifelong, long-term screening adherence, rather than one-time compliance. This is especially important because CRC screening can be unpleasant and if individuals are not clear of their risk and other important information about CRC, they may be reluctant to continue with a screening program. Having at least one first-degree relative (FDR) with CRC increases an individual's risk of developing the disease. Many relatives of CRC probands are ineligible for genetic testing and, therefore, do not receive information from a healthcare provider about the disease. Providing relatives of CRC probands with information about their risk of developing CRC, screening information, and other CRC-related health information, may increase knowledge and screening compliance as has been shown in relatives of breast cancer patients. Previous educational interventions with relatives of breast cancer probands have demonstrated increased knowledge, screening behaviour, risk comprehension, and decreased distress. While these interventions have been effective with relatives of breast cancer patients, these interventions have not been conducted to date with relatives of CRC patients. We believe that relatives of CRC patients could also benefit from this type of educational session. Educational interventions with relatives of breasts cancer patients have been conducted in-person, however in clinical genetic counseling, sessions are conducted both in-person and by telephone. Telephone counseling has become widespread in clinical services despite a lack of evidence to support its effectiveness compared to in-person counseling. Preliminary studies have shown that telephone interventions increase participation in screening programs, but few studies have directly compared telephone and in-person counseling. The primary aim of this study is to test the efficacy of two modes (in-person vs. telephone) of providing a risk counseling and health promotion intervention for relatives of CRC probands on measures of knowledge of CRC risk and health-related factors, comprehension of risk, understanding of screening recommendations and intent to adopt an appropriate screening regimen. Participants will be randomized into one of three study arms (in-person, telephone, control). An assessment pre- and post- intervention will be conducted. In addition, longer-term follow-ups will be carried out two months and one year following the intervention to examine the sustainability of the intervention effect.

ELIGIBILITY:
Inclusion Criteria:

* at least one First Degree Relative (FDR) with Colorectal Cancer
* be between the ages of 25 and 65 years
* live within one hour of Toronto

Exclusion Criteria:

* previous diagnosis of Colorectal Cancer or other malignancy
* family history suggestive of hereditary Colorectal Cancer
* history of major psychiatric disorder (i.e. schizophrenia, active psychosis, major depression)
* failure to provide consent.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Colorectal cancer risk comprehension and screening knowledge | 1 year
Intent to screen the colon | 1 year
Colon screening behaviour | 2 years

SECONDARY OUTCOMES:
Personality | Baseline
Psychosocial functioning | 1 year
Satisfaction | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Esplen, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Health Sciences Centre, Memorial University, St. John's, Newfoundland and Labrador
  - University Health Network, Toronto, Ontario